CLINICAL TRIAL: NCT03967873
Title: Prevalence of Preoperative Short-acting Mimetic beta2 Therapy by Parents of Asthmatic Children Attending Emergency Room for Asthma Attack
Brief Title: Child Asthma : What Parents Attitude During an Asthma Attack at Home Before Consulting the Pediatric Emergencies
Acronym: ASPECT
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ASPECT (29BRC18.0201)
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Asthma in Children; Asthma Attack; Therapeutic Adherence
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
prospective multicenter observational study. Parents whose children meet the inclusion criteria complete a questionnaire assessing the child's follow-up, the management of the current asthma attack, and the treatment provided at home.

The main objective is to calculate the prevalence of placement of short-acting bronchodilators. The secondary objectives are to describe the factors associated with their implementation.

ELIGIBILITY:
Inclusion Criteria:

* child over 2 years emergency room consultant for asthma attack
* child whose parents did not express their opposition to participate and completed the non-objection form
* child consultant in pediatric emergencies of Quimper and Brest

Exclusion Criteria:

* child whose age is not between 2 and 15 years old
* cough equivalent of asthma
* history of cardiac or pulmonary pathology or prematurity
* refusal to participate

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children between 2 and 15 years old in Quimper or Brest emergency department for asthma attacks whose parents agree to fill in a questionnaire about their pre-hospital attitude.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
prevalence of short-acting bronchodilator induction in children attending emergency room for asthma attack | 1 hour

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Brest, Brest
  - Ch Quimper, Quimper